CLINICAL TRIAL: NCT06739707
Title: A Multiple Dose, Randomized, Placebo-controlled, Dose-escalating Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Subcutaneously Administered MD-18 for Healthy Subjects With Overweight or Obesity
Brief Title: Subcutaneously Administered MD-18 for the Treatment of Obesity and Diabetes
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Cohen Global, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: MD-18-02
Record Dates: First submitted 2024-12-04; First posted 2024-12-18 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-02

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Intervention Model Description: Dosing will be in 7 dose cohorts. Cohorts 1 through 6 will be comprised of six subjects in each cohort using 4:2 (active: placebo) randomization. Thus, there will be four subjects receiving drug and two receiving placebo in each cohort. Cohort 7 will comprise 18 Obese subjects, in which 12 subjects will receive MD-18 and six will receive placebo. A total of 54 subjects will be enrolled in this study, with 36 receiving MD-18 and 18 receiving placebo. There is no need to wait for the completion of one cohort (Day 28) before proceeding to the next. Once all subjects for Cohort 1 have been recruited, the site should begin recruitment for Cohort 2, even while Cohort 1 is still ongoing. This process should continue for subsequent cohorts.
  The highest dose that is safe and tolerable in all subjects will be determined as the Maximum Tolerable Dose .
Who Masked: Participant, Investigator
Masking Description: Study medication will be supplied in labelled vials,clearly identifying the contents and indicating that the product is an investigational drug. An unblinding pharmacist at the clinical site will be responsible for the appropriate amount of vials to be dispnsed to each subject according to the randomization scheme. A blinded nurse will draw the correct amount of study medication into a syringe based on the subject's assigned arm, and administer the injection to the subject.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- A dose of 74 mg of MD-18 or placebo three times per week for 4 consecutive weeks (Experimental): Cohort 1: Four subjects will be administered a dose of 74 mg of MD-18 and two will receive placebo subcutaneously three times per week for 4 consecutive weeks
  Interventions: Drug: MD-18; Drug: Placebo
- A dose of 114 mg of MD-18 or placebo three times per week for 4 consecutive weeks (Experimental): Cohort 2: Four subjects will be administered a dose of 114 mg of MD-18 and two will receive placebo subcutaneously three times per week for 4 consecutive weeks.
  Interventions: Drug: MD-18; Drug: Placebo
- A dose of 227 mg of MD-18 or placebo three times per week for 4 consecutive weeks (Experimental): Cohort 3: Four subjects will be administered a dose of 227 mg of MD-18 and two will receive placebo subcutaneously three times per week for 4 consecutive weeks.
  Interventions: Drug: MD-18; Drug: Placebo
- A weekly dose of 302 mg of MD-18 or placebo for 4 consecutive weeks (Experimental): Cohort 4: Four subjects will be administered a weekly dose of 302 MD-18 and two will receive placebo subcutaneously for 4 consecutive weeks.
  Interventions: Drug: MD-18; Drug: Placebo
- A dose of 302 mg of MD-18 or placebo three times per week for 4 consecutive weeks (Experimental): Cohort 5: Four subjects will be administered a dose of 302 mg of MD-18 and two will receive placebo subcutaneously three times per week for 4 consecutive weeks.
  Interventions: Drug: MD-18; Drug: Placebo
- A daily dose of 302 mg of MD-18 or placebo for 4 consecutive weeks (Experimental): Cohort 6: Four subjects will be administered a daily dose of 302 mg of MD-18 and two will receive placebo subcutaneously for 4 consecutive weeks.
  Interventions: Drug: MD-18; Drug: Placebo
- The highest tolerated dose/dose-frequency identified in the first six cohorts (Experimental): Cohort 7: Twelve non-diabetic obese subjects will be treated with the highest tolerated dose/dose-frequency identified in the first six cohorts and six subjects will be administered placebo.
  Interventions: Drug: MD-18; Drug: Placebo

INTERVENTIONS:
Drug: MD-18 — MD-18 administered subcutaneously to healthy individuals with overweight or obesity.
Drug: Placebo — Placebo administered subcutaneously to healthy individuals with overweight or obesity.

SUMMARY:
A Multiple Dose, Randomized, Placebo-controlled, Dose-escalating Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Subcutaneously Administered MD-18 for healthy subjects with overweight or obesity

DETAILED DESCRIPTION:
This study will be conducted as a single center study, at the Sheba Medical Center, Israel. Escalating daily doses of MD-18 or placebo will be administered subcutaneously to each subject over a 4-week period with a 7-day follow-up period. 54 patients will be enrolled across 7 cohorts. Each of the cohorts will enroll 4 active and two placebo subjects, except for the final cohort. Cohort 7 will be comprised of obese subjects and will enroll 12 active and 6 placebo subjects. Starting dose has been determined from the SAD study (CG MD-18-01). Cohorts will receive 74 mg MD-18 three times weekly, (starting dose), 114 mg three times weekly, 227 mg three times weekly, 302 mg once weekly, 302 mg three times weekly or 302 mg daily using 4:2 (active:placebo) randomization; all doses refer to the MD-18 salt. A total of 36 subjects will receive active therapy across seven cohorts (24 in the first six cohorts and 12 in the seventh cohort) and 18 subjects will receive placebo. The study will be conducted on an outpatient basis, with visits performed as shown in the schedule of events.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 18-70 years, both genders.
2. BMI:

   * Cohorts 1-6: 25-34.9
   * Cohort 7: 30.0-44.9
3. HbA1c <6.5%
4. Healthy as determined by a physician, based on history, medical examination, vital signs, laboratory tests, cardiac monitoring and respiratory function. History must comply with the following:

   1. Absence of clinically significant illness or major surgery within the preceding 12 weeks.
   2. Absence of clinically significant history of neurological, endocrine, cardiovascular, pulmonary, hematological, immunologic, psychiatric, gastrointestinal, renal, hepatic, and/or metabolic disease as per PI decision.
5. Male subjects with female partners of childbearing potential must agree to utilize an approved contraceptive during the study.
6. Female subjects of child-bearing potential with negative urine pregnancy test at screening and who agree to use contraception during the study.
7. Female subjects of non-child-bearing potential (i.e. tubal ligation, hysterectomy, or postmenopausal).
8. Subjects must provide written informed consent and be willing and able to comply with study procedures.

Exclusion Criteria:

1. History of excessive alcohol use (defined as >21 drinks per week for males and >14 drinks per week for females), recreational drug use within the past three months, or failure on urinary drug screen. Note: use of Cannabinoids for medical purposes is allowed.
2. Pregnant or breastfeeding within six months of screening assessment.
3. Substantial changes in eating habits or exercise routine within the preceding three months.
4. Evidence of eating disorders.
5. >5% weight change in the past three months.
6. Bariatric surgery within the past five years.
7. Moderate renal impairment ( Glomerular filtration rate<60 mg/mL/1.73m2)
8. Liver function tests greater than twice the upper limit of normal upon repeated measurements.
9. Diseases interfering with metabolism and or ingestive behavior (e.g., myxedema, Cushing's disease, schizophrenia, major psychoses, unmanaged depression).
10. Use of medications affecting body weight within the past three months, unless on a stable dose, with weight stability in the preceding three months. These medications include:

    1. Drugs approved for the treatment of obesity
    2. Cyproheptadine or medroxyprogesterone
    3. Atypical anti-psychotic drugs
    4. Tricyclic antidepressants
    5. Lithium, MAO's, glucocorticoids
    6. SSRIs or SNRIs
    7. Anti-epileptic drugs
11. Any clinically significant abnormality following the Investigator's review of the physical examination and clinical laboratory tests.
12. A baseline (screening echocardiogram result) prolongation of ventricular activation and recovery interval after repeated measurements of >450 milliseconds; a history of unexplained syncope, cardiac arrest, unexplained cardiac arrhythmias or torsades de pointes, structural heart disease, or a family history of Long QT Syndrome.
13. Use drugs of abuse within the preceding three months.
14. The last dose of an investigational drug in other clinical trial was within the month prior to dosing in the present study. Note: Volunteers from the previous Phase 1a trial (MD-18-01) may be recruited for the current study, provided that at least 12 weeks have passed since their last dose of the investigational product.
15. A positive result for any of the following tests: hepatitis B virus (HBV), hepatitis C virus (HCV), human immunodeficiency viruses (HIV) and Treponema pallidum.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
To determine the safety and tolerability multiple subcutaneous doses of MD-18 in overweight or obese but otherwise healthy subjects, as assessed by the collection of Adverse events. | Through study completion, an average of 8 months
  All adverse events, exacerbations of concomitant illnesses, or events known to be related to underlying disease processes or concomitant medications are to be recorded on the case report form throughout the study. Should there be more than 2 subjects receiving MD-18 with an adverse event grade 4 or 5 that is at least possibly related to MD-18, the study will be put on immediate hold and the data will be reviewed by the site Principal Investigator (PI) and the company Chief Medical Officer (CMO) before proceeding.
To determine the safety and tolerability multiple subcutaneous doses of MD-18 in overweight or obese but otherwise healthy subjects, as assessed by the collection of body temperature. | During the following study visits: Screening, Day 1,7,14,21,28 and 35) and at the study visits of the 8 weeks study extension period on days 42,56,70,84 and 92 (Only for subjects that have agreed to participate from Cohort 7)
  Body temperature measurements in Celsius (°C) will be conllected at the visits specified in the study protocol's Schedule of Events. If any clinically significant findings or machine/equipment errors occur, the measurement will be repeated. Any confirmed clinically significant result will be recorded as adverse events (AEs).
To determine the safety and tolerability multiple subcutaneous doses of MD-18 in overweight or obese but otherwise healthy subjects, as assessed by the collection of Serum chemistry. | During the screening visit, Day 1, 7,28,35 and at the study visits of Day 56,84 and 92 at the 8 weeks study extension period (Only for subjects that have agreed to participate from Cohort 7).
  Collection of blood samples for serum chemistry
To determine the safety and tolerability multiple subcutaneous doses of MD-18 in overweight or obese but otherwise healthy subjects, as assessed by the collection of body weight | During each study visit and at the study visits of the 8 weeks study extension period (Only for subjects that have agreed to participate from Cohort 7)
  Body weight (in kilograms) will be measured. To ensure consistency and accuracy, all subjects will be measured while wearing only undergarments or light clothing, without shoes. A calibrated scale will be used consistently throughout the study. In addition, weight measurements along with the screening height measurement will be combined to report BMI in kg/m^2
To determine the safety and tolerability multiple subcutaneous doses of MD-18 in overweight or obese but otherwise healthy subjects, as assessed by the collection of Electrocardiogram examination. | at screening (visit 1; Day -7) and days 7, 28 and 35. On Day 92 (for the 8 weeks extension period Only for subjects that have agreed to participate from Cohort 7).
  12-lead triplicate ECGs will be obtained.
  The ECG machine will automatically calculate the following:
  Heart rate ( refers to the number of contractions of the heart per minute) PR interval (PR interval is the time from the beginning of the P wave (atrial depolarization) to the beginning of the QRS complex.
  QRS complex (represents the depolarization of ventricles And the beginning of systole and ventricular contraction).
  QT interval (is the time from the beginning of the QRS complex, representing ventricular depolarization, to the end of the T wave, resulting from ventricular repolarization).
  QTc interval (is the QT interval corrected for heart rate).
To determine the safety and tolerability multiple subcutaneous doses of MD-18 in overweight or obese but otherwise healthy subjects, as assessed by the collection of respiration rate | During the following study visits: Screening, Day 1,7,14,21,28 and 35) and at the study visits of the 8 weeks study extension period on days 42,56,70,84 and 92 (Only for subjects that have agreed to participate from Cohort 7)
  Respiration rate in breaths per minute will be collected at the visits specified in the study protocol's Schedule of Events. If any clinically significant findings or machine/equipment errors occur, the measurement will be repeated. Any confirmed clinically significant result will be recorded as adverse events.
To determine the safety and tolerability multiple subcutaneous doses of MD-18 in overweight or obese but otherwise healthy subjects, as assessed by the collection of heart rate | During the following study visits: Screening, Day 1,7,14,21,28 and 35) and at the study visits of the 8 weeks study extension period on days 42,56,70,84 and 92 (Only for subjects that have agreed to participate from Cohort 7)
  Heart rate in beats per minute will be collected at the visits specified in the study protocol's Schedule of Events. If any clinically significant findings or machine/equipment errors occur, the measurement will be repeated. Any confirmed clinically significant result will be recorded as adverse events.
To determine the safety and tolerability multiple subcutaneous doses of MD-18 in overweight or obese but otherwise healthy subjects, as assessed by the collection of systolic and diastolic blood pressure | During the following study visits: Screening, Day 1,7,14,21,28 and 35) and at the study visits of the 8 weeks study extension period on days 42,56,70,84 and 92 (Only for subjects that have agreed to participate from Cohort 7)
  Systolic and diastolic blood pressure in millimeters of mercury (mmHg) will be collected at the visits specified in the study protocol's Schedule of Events. If any clinically significant findings or machine/equipment errors occur, the measurement will be repeated. Any confirmed clinically significant result will be recorded as adverse events.
To determine the safety and tolerability multiple subcutaneous doses of MD-18 in overweight or obese but otherwise healthy subjects, as assessed by the collection of Hematology blood test | During the screening visit, Day 1, 7,28,35 and at the study visits of Day 56,84 and 92 at the 8 weeks study extension period (Only for subjects that have agreed to participate from Cohort 7).
  Collection of Hematology blood test
To determine the safety and tolerability multiple subcutaneous doses of MD-18 in overweight or obese but otherwise healthy subjects, as assessed by the collection of coagulation panel | During the screening visit, Day 1, 7,28,35 and at the study visits of Day 56,84 and 92 at the 8 weeks study extension period (Only for subjects that have agreed to participate from Cohort 7).
  Collection of blood samples for coagulation panel.
To determine the safety and tolerability multiple subcutaneous doses of MD-18 in overweight or obese but otherwise healthy subjects, as assessed by the collection of Urine analysis | During the screening visit, Day 1, 7,28,35 and at the study visits of Day 56,84 and 92 at the 8 weeks study extension period (Only for subjects that have agreed to participate from Cohort 7).
  Collection of urine samples for Urine analysis
To determine the safety and tolerability multiple subcutaneous doses of MD-18 in overweight or obese but otherwise healthy subjects, as assessed by the collection of height | At the study screening visit (Day -28 to day -1 Pre-Treatment)
  Height (in centimeters) will be collected only at the screening visit and will be combined with the body weight measurements in order to calculate the body mass index (BMI) in kg/m2. A calibrated scale will be used consistently throughout the study.

SECONDARY OUTCOMES:
To determine the safety and tolerability multiple subcutaneous doses of MD-18 in overweight or obese but otherwise healthy subjects, as assessed by the collection of pharmacokinetic for Area Under the Curve (AUC) analysis | Before dose administration and at 0.5, 1, 2, 4, and 8 hours after dose administration on Days 1 and 28 of each dose level.
  Plasma samples will be collected for the pharmacokinetic analysis of Area Under the Curve (AUC) for various time intervals: AUC0-1h, AUC0-2h, AUC0-4h, AUC0-12h, AUC0-24h, and AUCinf.
  Pharmacokinetic parameters will be summarized using descriptive statistics at each scheduled assessment time point.
To determine the safety and tolerability multiple subcutaneous doses of MD-18 in overweight or obese but otherwise healthy subjects, as assessed by the collection of pharmacokinetic for Maximum concentration of MD-18 (Cmax) analysis | Before dose administration and at 0.5, 1, 2, 4, and 8 hours after dose administration on Days 1 and 28 of each dose level.
  Plasma samples will be collected for the pharmacokinetic analysis of Maximum concentration of MD-18 (Cmax).
To determine the safety and tolerability multiple subcutaneous doses of MD-18 in overweight or obese but otherwise healthy subjects, as assessed by the collection of pharmacokinetic for Minimum concentration of MD-18 between doses (Cmin) analysis | Before dose administration and at 0.5, 1, 2, 4, and 8 hours after dose administration on Days 1 and 28 of each dose level.
  Plasma samples will be collected for the pharmacokinetic analysis of inimum concentration of MD-18 between doses (Cmin).
  Pharmacokinetic parameters will be summarized using descriptive statistics at each scheduled assessment time point.
To determine the safety and tolerability multiple subcutaneous doses of MD-18 in overweight or obese but otherwise healthy subjects, as assessed by the collection of Plasma samples for the pharmacokinetics analysis of Time to reach maximum concentration | Before dose administration and at 0.5, 1, 2, 4, and 8 hours after dose administration on Days 1 and 28 of each dose level.
  Plasma samples will be collected for the pharmacokinetic analysis of Time to reach maximum concentration of MD-18 (Tmax).
  Pharmacokinetic parameters will be summarized using descriptive statistics at each scheduled assessment time point.
To determine the safety and tolerability multiple subcutaneous doses of MD-18 in overweight or obese but otherwise healthy subjects, as assessed by the collection of pharmacokinetic for the analysis of Half-life (t½) | Before dose administration and at 0.5, 1, 2, 4, and 8 hours after dose administration on Days 1 and 28 of each dose level.
  Plasma samples will be collected for the pharmacokinetic analysis of the study drug MD-18 Half-life (t½).
  Pharmacokinetic parameters will be summarized using descriptive statistics at each scheduled assessment time point.
To determine the safety and tolerability multiple subcutaneous doses of MD-18 in overweight or obese but otherwise healthy subjects, as assessed by the collection of Plasma samples for pharmacokinetics analysis of clearance rate (CL/F) | Before dose administration and at 0.5, 1, 2, 4, and 8 hours after dose administration on Days 1 and 28 of each dose level.
  Plasma samples will be collected for the pharmacokinetic analysis of the study drug MD-18 clearance rate (CL/F).
  Pharmacokinetic parameters will be summarized using descriptive statistics at each scheduled assessment time point.
To determine the safety and tolerability multiple subcutaneous doses of MD-18 in overweight or obese but otherwise healthy subjects, as assessed by the collection of Plasma samples for the pharmacokinetics analysis of volume of distribution (V/F) | Before dose administration and at 0.5, 1, 2, 4, and 8 hours after dose administration on Days 1 and 28 of each dose level.
  Plasma samples will be collected for the pharmacokinetic analysis of the study drug MD-18 volume of distribution (V/F).
  Pharmacokinetic parameters will be summarized using descriptive statistics at each scheduled assessment time point.

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Please Select, Israel

IPD SHARING:
Plan to Share IPD: Undecided